CLINICAL TRIAL: NCT00694772
Title: Coblation-Tonsillotomy Versus Electrocautery-Tonsillectomy for Treatment of Moderate and Severe Obstructive Sleep Apnea in Children: A Randomized, Prospective, Single-Blinded Study
Brief Title: Coblation-Tonsillotomy vs Electrocautery-Tonsillectomy for the Treatment of Obstructive Sleep Apnea (OSA) in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: ArthroCare Corporation (Other); Calgary Health Region (Other)
Responsible Party: Derek Drummond, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E-21417
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2008-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; OSA; Apnea hypopnea index; AHI; Coblation; Electrocautery; Tonsillectomy; Tonsillotomy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electrocautery (Active Comparator)
  Interventions: Procedure: Electrocautery-tonsillectomy
- Coblation (Experimental)
  Interventions: Procedure: Coblation-tonsillotomy

INTERVENTIONS:
Procedure: Electrocautery-tonsillectomy — standard of care electrocautery tonsillectomy
  Arms: Electrocautery
Procedure: Coblation-tonsillotomy — use of Arthrocare Coblation Technology to perform tonsillotomy
  Other Names: alternative procedure name: subcapsular tonsillectomy
  Arms: Coblation

SUMMARY:
Removal of the adenoid and tonsils, known as an adenotonsillectomy (AT) is one of the most frequently performed surgical procedures in North America. The two most prevalent indications for this procedure in children are recurrent bacterial tonsillitis and obstructive sleep apnea (OSA). OSA is a common childhood condition that is characterized by upper airway obstruction, disturbed sleep and disrupted normal respiratory gas exchange. In the majority of children with OSA, overgrowth of the adenoid and tonsils is the primary underlying aetiology, making tissue removal via AT the standard of care. The purpose of this study is to evaluate the effectiveness of two different surgical techniques, electrocautery-tonsillectomy and coblation-tonsillotomy, in the treatment of obstructive sleep apnea (OSA) in children.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe OSA on PSG (AHI ≥ 5.0)
* Pronounced tonsillar hyperplasia on physical exam
* No previous tonsil or adenoid surgery
* No history of recurrent tonsillitis
* Participants and their families must be willing to comply with follow-up
* Parents/caregivers fluent in English

Exclusion Criteria:

* Severe co-morbidities, including, but not limited to, poorly controlled asthma, chromosomal abnormalities, and developmental delay

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2008-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Compare coblation-tonsillotomy to electrocautery-tonsillectomy as a treatment of obstructive sleep apnea (OSA), as assessed by apnea-hypopnea index (AHI) measured on polysomnography (PSG) | 6 months and 2 years post-op

SECONDARY OUTCOMES:
Evaluate post-operative pain and analgesic use associated with electrocautery-tonsillectomy and coblation-tonsillotomy | 1 week post-op
Evaluate quality of life following coblation-tonsillotomy and electrocautery-tonsillectomy for the treatment of OSA | 6-8 weeks post-op

CONTACTS AND LOCATIONS:
Overall Officials: Derek S Drummond, MD, MPH, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada